CLINICAL TRIAL: NCT04262791
Title: A Multicenter, Non-Drug Interventional Study for the Technical Development and Validation of the Nocturnal Scratch Algorithm for Use in Future Programs
Brief Title: A Non-Drug Study Detecting And Quantifying Nocturnal Scratch Behaviors From Wrist Actigraphy Data In Adult Healthy Volunteers And Participants With Atopic Dermatitis (AD)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Strategic Considerations
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: F20-093
Record Dates: First submitted 2020-02-07; First posted 2020-02-10 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2022-02

CONDITIONS: Atopic Dermatitis
Keywords: Nocturnal Scratch Algorithm; Atopic Dermatitis (AD); Wrist Actigraphy
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Healthy Volunteers (Experimental): Healthy participants will be monitored overnight for two consecutive nights at an inpatient setting to collect wrist actigraphy and videography data. Sleep headband (at sites where polysomnography (PSG) is available and performed) data will be collected on Night 2.
  Interventions: Device: Wrist Actigraphy Device; Device: Sleep Headband
- Participants With Atopic Dermatitis (AD) (Experimental): Participants with AD will be monitored overnight for two consecutive nights at an inpatient setting to collect wrist actigraphy and videography data. Sleep headband (at sites where polysomnography (PSG) is available and performed) data will be collected on Night 2. Participants will also be monitored at home via wrist actigraphy, sleep headband when available in the outpatient setting for 7 consecutive nights.
  Interventions: Device: Wrist Actigraphy Device; Device: Sleep Headband

INTERVENTIONS:
Device: Wrist Actigraphy Device — Wrist Actigraphy Device
Device: Sleep Headband — Sleep Headband
  Other Names: Dreem 2 Headband

SUMMARY:
Sleep disturbance is very common in patients with atopic dermatitis (AD) and is a major factor leading to impaired quality of life. Nocturnal scratching is one of the factors causing sleep disturbance in AD patients. This study aims to develop and validate a digital algorithm for accurately and reliably detecting and quantifying nocturnal scratch behaviors related to AD using wrist actigraphy data.

Wrist actigraphy is an investigational device being developed to detect and quantify scratching behaviors in patients with AD. This study will be conducted in 2 sequential stages: In Stage 1, an algorithm will be developed and in Stage 2 the algorithm developed will be validated. Adult healthy volunteers or participants with AD will be enrolled. Approximately 14 healthy volunteers, 14 AD patients with low disease activity and 28 AD patients with high disease activity will be enrolled in the study in 5 sites across the United States.

No drug will be administered as a part of this study.

Participants enrolled in this study may experience discomfort or inconvenience related to the study procedures. Participants will be enrolled and monitored overnight for two consecutive nights at an inpatient setting at a hospital or clinic. The impact of nocturnal scratching on sleep parameters will be assessed by videography, actigraphy, sleep headband and completing questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers in general good health with no diagnosis of AD or any other dermatologic disorder that interferes with study assessments.
* For subjects with AD:
* Chronic AD with onset of symptoms at least 1 year prior to Day 1 and participant meets American Academy of Dermatology (AAD) criteria.
* Participant meets all of the following disease activity criteria:

  * For AD subjects with high disease activity (AD-High):

    * Pruritus over the last 7 days (numerical rating scale 7-Day version [NRS-7]) >= 4 at the Screening and Day 1 visits.
    * At least one of the following:

      * Eczema Area and Severity Index (EASI) score > 7 at the Screening and Day 1 visits; OR
      * Validated Investigator Global Assessment for AD (vIGA-AD) score >= 3 at the Screening and Day 1 visits;
  * For AD subjects with low disease activity (AD-Low):

    * Pruritus over the last 7 days (NRS-7) >= 2 at the Screening and Day 1 visits.
    * Does not meet AD-High criteria as described.
    * Satisfy at least one of the following:

      * EASI score >= 3 at the Screening and Day 1 visits OR
      * vIGA-AD score >= 1 at the Screening and Day 1 visits.

Exclusion Criteria:

* Significant eczema on wrists where devices will be worn that, in the opinion of the participant or investigator would likely lead to non-compliance.
* Interference (e.g., hairstyle) with the ability of Dreem 2 headband to collect sensor data.
* Unstable medical disorder or other condition that in the investigator's opinion may interfere with study procedures or study objectives.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2020-02-17 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Total Scratch Duration Per Night | Up to 10 Days
  Total scratch duration per night (seconds/night) is measured by actigraphy and videography.

SECONDARY OUTCOMES:
Number of Scratching Events | Up to 10 Days
  Number of scratching events are measured by actigraphy and videography
Scratch Rate | Up to 10 Days
  Scratch rate is measured by actigraphy.
Scratch Duration | Up to 10 Days
  Scratch duration is defined as percentage of total rest/sleep time as measured by actigraphy and videography
Comparison of Actigraphy-Based Scratches to Videography-Based Scratches | Up to 10 Days
  Actigraphy-based scratches, as determined by the final algorithm determined in Stage 1, will be compared to videography-based scratches over epoch in which scratch is scored by either actigraphy or videography (and ignoring epochs in which no scratch is scored by either method) over the sleep period.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (3):
- United States (3):
  - PPD Clinical Research Unit /ID# 217010, Orlando, Florida
  - Acpru /Id# 217345, Grayslake, Illinois
  - Univ Rochester Med Ctr /ID# 217490, Rochester, New York

IPD SHARING:
Plan to Share IPD: No